CLINICAL TRIAL: NCT05712434
Title: A Multi-center, Stepped-wedge, Cluster-randomized Control Trial to Evaluation the Effectiveness of Chlorhexidine to Prevent Catheter-associated Urinary Tract Infection
Brief Title: Chlorhexidine to Prevent Catheter-related Urinary Tract Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other); Hualien Tzu Chi General Hospital (Other); National Taiwan University Hospital Hsin-Chu Branch (Other); Lotung Poh-Ai Hospital (Other); Min-Sheng General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 202212030MIFA
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2023-01

CONDITIONS: Urinary Tract Infections
Keywords: chlorhexidine; catheter-related urinary tract infection; disinfection; bundle care; Foley catheter; urinary catheter
MeSH Terms: conditions — Urinary Tract Infections | interventions — Chromogranins

STUDY DESIGN:
Intervention Model Description: Each enrolled units will start with iodine protocol, and then switched to CHG protocol at designated time, followed by CHG plus protocol subsequently. Each unit will be randomized in to three different groups (A, B, and C):
  Group A) 2 months of iodine protocol, followed by 4 months of CHG protocol, followed by 6 months of CHG plus protocol.
  Group B) 4 months of iodine protocol, followed by 4 months of CHG protocol, followed by 4 months of CHG plus protocol.
  Group C) 6 months of iodine protocol, followed by 4 months of CHG protocol, followed by 2 months of CHG plus protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Long CHG Intervention (Experimental): 2 months of iodine protocol, followed by 4 months of CHG protocol, followed by 6 months of CHG plus protocol.
  Interventions: Other: Long Intervention
- Mid-length CHG Intervention (Experimental): 4 months of iodine protocol, followed by 4 months of CHG protocol, followed by 4 months of CHG plus protocol.
  Interventions: Other: Mid-length Intervention
- Short CHG Intervention (Experimental): 6 months of iodine protocol, followed by 4 months of CHG protocol, followed by 2 months of CHG plus protocol.
  Interventions: Other: Short Intervention

INTERVENTIONS:
Other: Long Intervention — Each unit will start with iodine protocol, which uses 10% povidone-iodine for disinfection during Foley insertion, for 2 months. After the designated duration of protocol (determined by the results of randomization), each unit will than switched to CHG protocol for 4 months, in which 2% aqueous chlorhexidine solution are used instead of iodine solution. Subsequently, in the final 6-month phase of study, each unit will than switched to CHG plus protocol, in which 0.05% CHG impregnated gel will be used alongside 2% CHG solution during Foley insertion.
  Other Names: 4-month CHG and 6-month CHG plus
  Arms: Long CHG Intervention
Other: Mid-length Intervention — Each unit will start with iodine protocol, which uses 10% povidone-iodine for disinfection during Foley insertion, for 4 months. After the designated duration of protocol (determined by the results of randomization), each unit will than switched to CHG protocol for 4 months, in which 2% aqueous chlorhexidine solution are used instead of iodine solution. Subsequently, in the final 4-month phase of study, each unit will than switched to CHG plus protocol, in which 0.05% CHG impregnated gel will be used alongside 2% CHG solution during Foley insertion.
  Other Names: 4-month CHG and 4-month CHG plus
  Arms: Mid-length CHG Intervention
Other: Short Intervention — Each unit will start with iodine protocol, which uses 10% povidone-iodine for disinfection during Foley insertion, for 6 months. After the designated duration of protocol (determined by the results of randomization), each unit will than switched to CHG protocol for 4 months, in which 2% aqueous chlorhexidine solution are used instead of iodine solution. Subsequently, in the final 2-month phase of study, each unit will than switched to CHG plus protocol, in which 0.05% CHG impregnated gel will be used alongside 2% CHG solution during Foley insertion.
  Other Names: 4-month CHG and 2-month CHG plus
  Arms: Short CHG Intervention

SUMMARY:
The study is to investigate whether chlorhexidine (CHG)-based antiseptics is more effective to prevent catheter-related urinary tract infection (CAUTI) among inhospital patients who required Foley catheter insertion. This is a cluster-randomised, step-wedged clinical trial, in which every participated unit will used three different Foley catheter insertion protocols during the study period:

1. Iodine protocol: using 10% povidone-iodine as the primary antiseptic during Foley insertion. This is the routine practice before this study in the participated hospital, as well as many Taiwanese hospitals.
2. CHG protocol: instead of povidone-iodine solution, use 2% aqueous CHG solution as the primary disinfectant during Foley solution.
3. CHG plus protocol: additional to 2% CHG solution, added 0.5% CHG impregnated gel as the lubrication during Foley insertion.

DETAILED DESCRIPTION:
This is a open-labelled, cluster-randomized, step-wedged clinical trial aimed to observe the incidence if CAUTI during the designated study period (12 months for all participated units). All included units will start with the iodine protocol, which is the standard practice in the hospital, and then switched to CHG protocol than CHG plus protocol according to the results of randomization. Each unit will be randomized in to three different groups (A, B, and C):

Group A) 2 months of iodine protocol, followed by 4 months of CHG protocol, followed by 6 months of CHG plus protocol.

Group B) 4 months of iodine protocol, followed by 4 months of CHG protocol, followed by 4 months of CHG plus protocol.

Group C) 6 months of iodine protocol, followed by 4 months of CHG protocol, followed by 2 months of CHG plus protocol.

All unit will be monitored and compared for the occurrence of CAUTI, which is defined in accordance to the definition from the National Healthcare Safety Network (USCDC).

ELIGIBILITY:
This is a cluster-randomized clinical trial. The enrollment is for healthcare units (wards, ICUs) in the participated hospitals rather than individuals. Patients who were admitted in the included unit with be enrolled in our study automatically.

Inclusion Criteria (for units):

* Adult acute care wards or intensive care units, which primarily care for adult patients aged above 18 years.
* Currently not using chlorhexidine as disinfectants for Foley catheter insertion or routine care.
* Had patients who required Foley catheter insertion during the last 12 months prior to inclusion.
* Willing to implant measures to improve the rate of CAUTI, and to participate and follow the study protocol in our study.

Exclusion Criteria (for units):

* Units currently using chlorhexidine as disinfectants for Foley catheter insertion or routine care.
* Wards or intensive care units with patients aged below 18 years of age in their routine practice.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30994 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of catheter-related urinary tract infection | During the entire observation period (12 months)
  The incidence of CAUTI, according to the updated definition of National Healthcare Safety Network (any Candida species will be excluded as pathogen)

SECONDARY OUTCOMES:
Incidence of catheter-related urinary tract infection (including candiduria) | During the entire observation period (12 months)
  The incidence of CAUTI, according to the updated definition of National Healthcare Safety Network, but candiduria not excluded as pathogen
Incidence of catheter-related urinary tract infection, by different clinical relevant isolates | During the entire observation period (12 months)
  The incidence of CAUTI caused by different clinical relevant isolates (Pseudomonas aeruginosa, enterococci, enteric gram-negative bacteria, other pseudomonads, etc.)

OTHER OUTCOMES:
The occurrence of severe adverse effects related to topical CHG disinfection | During the entire observation period (12 months)
  The occurrence of severe adverse effects related to topical CHG disinfection

CONTACTS AND LOCATIONS:
Overall Officials: Yee-Chun Chen, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Owing to the study design, informed consent is waived by the Research Ethic Committee of National Taiwan University Hospital. Therefore, individual data could not be shared as there is no consent.